CLINICAL TRIAL: NCT00824278
Title: The Use of a Distress Thermometer in a Pediatric Research Setting: An Exploratory, Pilot Study
Brief Title: The Use of a Distress Thermometer in a Pediatric Research Setting: An Exploratory Pilot Study
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090022; 09-M-0022
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-05-31

CONDITIONS: Cancer; HIV Infections
Keywords: Pediatrics; Distresss Screening; Cancer; Neurofibromatosis; HIV; Pediatric Cancer; Distress Screening
MeSH Terms: conditions — Neoplasms; HIV Infections; Neurofibromatoses

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Medical illnesses and treatments can cause distress in patients, and medical professionals are very interested in identifying distress quickly to ensure that a patient can receive appropriate support and treatment. Adult patients often use a screening tool known as the Distress Thermometer to indicate the causes and levels of distress they feel. However, little work has been done on how to assess distress in pediatric patients. This study will investigate the effectiveness of the Distress Thermometer as a tool to accurately measure distress in pediatric patients, and determine whether primary caregivers and physicians can also use the Distress Thermometer to accurately gauge a patient s levels and sources of distress. The study will also investigate the effectiveness of the Distress Thermometer compared with other means of measuring fatigue, mood, and pain levels.

This study will include approximately 90 patients between 7 and 21 years of age who are currently enrolled in a National Institutes of Health pediatric research study. It will also include responses from the primary caregivers and primary medical providers of the patients involved in the study.

All patients will complete the Distress Thermometer s self-reported distress scale and other standardized measures of anxiety, depression, fatigue, and pain. In addition, patients between 18 and 21 years of age will be asked to assess the benefits and negative effects of participating in psychosocial research.

On the same day, the patient s primary caregiver and primary medical provider will complete a Distress Thermometer survey to estimate the patient s distress level. If either the patient or the primary caregiver indicate high levels of distress or mood symptoms, the researchers will offer them an opportunity to speak with a mental health professional. The primary medical provider will also receive a copy of the responses reported on the patient s Distress Thermometer.

DETAILED DESCRIPTION:
OBJECTIVE:

The purpose of this protocol is to evaluate a measure that would assist clinicians in assessing the presence of psychological distress in children and adolescents with serious medical illnesses.

Aim 1: To assess the inter-rater reliability of the Distress Thermometer by comparing ratings of the patient s distress given by the patient, the primary caregiver and the patient s primary medical provider.

Aim 2: To assess the concurrent validity (i.e. the extent to which a test correlates with other previously validated measures of similar constructs) of the Distress Thermometer, a brief screening tool for psychological distress, as compared to validated measures of psychological symptoms (i.e. depression, anxiety, pain and fatigue) in patients with pediatric cancer, Neurofibromatosis Type 1 (NF1) HIV-1 infection, Primary Immune Deficiencies (PIDs), DNA repair diseases, sickle cell disease, and Li-Fraumeni.

Aim 3: To assess the acceptability of completing the Distress Thermometer to patients, primary caregivers, and medical providers.

Aim 4: To assess the feasibility of administering the Distress Thermometer to patients with cancer, NF1, and HIV-1 infection, PIDs, and DNA repair diseases.

Secondary Aim 1: To assess the relationship between the caregiver s self-report of psychological symptoms and his or her rating of the patient s level of distress on the Distress Thermometer.

Secondary Aim 2: To assess whether patient ratings on the Distress Thermometer differ between the specific diseases, controlling for disease severity.

Secondary Aim 3: To assess the burden and benefits of participating in psychosocial research.

STUDY POPULATION:

This study is taking place at the National Institutes of Health (NIH) and Medstar Georgetown University Hospital. All outpatients, ages 7-21, enrolled in a research study either at the Pediatric Clinic, the Primary Immune Deficiency Clinic, or the Dermatology Clinic at the NIH with a diagnosis of pediatric cancer, NF-1, HIV, PIDs, and DNA repair, and those at risk for Li-Fraumeni (P53 positive)syndrome diseases will be invited to participate in this study. Additionally, all outpatients, ages 7-21, seen at Medstar Georgetown University Hospital for HIV or sickle cell disease will be invited to participate in this study.

DESIGN:

Each patient will complete a brief self-report distress scale (the Distress Thermometer) and standardized measures of depression, anxiety, pain, and fatigue. Additionally, all patients will be asked to assess the benefits and burdens of participating in psychosocial research.

Primary caregivers will rate their child s level of distress (using the Distress Thermometer), pain, fatigue anxiety and depression, and complete a self-report measure assessing their own psychological symptoms in addition to questions that assess the benefits and burdens of participating in psychosocial research.

The primary medical provider (physicians or nurse practitioners) will give their estimation of the patient s distress (using the Distress Thermometer).

All patients, primary caregivers and medical providers will assess the acceptability of completing the Distress Thermometer. Additionally, data collectors will assess the feasibility of administering the Distress Thermometer in a pediatric clinic. <TAB>

MEASURES:

Measures include the Distress Thermometer, a brief screening tool consisting of a single item rating of distress and a list of possible reasons for distress; the Children s Depression Inventory (CDI); the Brief Symptom Inventory 18 (BSI-18); the State Trait Anxiety Inventory (STAI); the Wong-Baker FACES Pain Scale; the Children s Fatigue Scales; an Acceptability and Feasibility scale for completion of the Distress Thermometer; and two questions regarding perception of research participation.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

* Age 7 to 21 years.
* Must be enrolled in a research protocol at the NIH or receiving medical treatment at Georgetown's Medical Center and be an outpatient at time of study. The treatment protocol PI will be contacted before a patient is approached to ensure that the patient is appropriate for enrollment into this protocol.
* Must have a parent/guardian available to complete the study measures.
* For patients less than 18 years of age, a legal guardian must provide informed consent and the patients must sign an assent document.
* Patients greater than or equal to 18 years of age must give informed consent and their parents need to sign the parent consent.
* Patients must speak English (as all instruments have not been validated in languages other than English.)

EXCLUSION CRITERIA:

- Presence of psychotic symptoms or cognitive impairment, which in the judgment of the Principal or Associate Investigator, or consulting psychiatrist would compromise the patient s ability to accurately complete the measures.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 289 (Actual)
Dates: Start 2009-01-13; Study Completion 2018-05-31

PRIMARY OUTCOMES:
Positive score on depression, anxiety, pain and fatigue measures.

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Allison TG, Williams DE, Miller TD, Patten CA, Bailey KR, Squires RW, Gau GT. Medical and economic costs of psychologic distress in patients with coronary artery disease. Mayo Clin Proc. 1995 Aug;70(8):734-42. doi: 10.4065/70.8.734. PMID 7630210
- [Background] Barton B, North K. Social skills of children with neurofibromatosis type 1. Dev Med Child Neurol. 2004 Aug;46(8):553-63. doi: 10.1017/s0012162204000921. PMID 15287247
- [Background] Battles HB, Wiener LS. From adolescence through young adulthood: psychosocial adjustment associated with long-term survival of HIV. J Adolesc Health. 2002 Mar;30(3):161-8. doi: 10.1016/s1054-139x(01)00341-x. PMID 11869922
- [Derived] Shain LM, Pao M, Tipton MV, Bedoya SZ, Kang SJ, Horowitz LM, Wiener L. Comparing Parent and Child Self-report Measures of the State-Trait Anxiety Inventory in Children and Adolescents with a Chronic Health Condition. J Clin Psychol Med Settings. 2020 Mar;27(1):173-181. doi: 10.1007/s10880-019-09631-5. PMID 31127422
- [Derived] Wiener L, Battles H, Zadeh S, Pao M. Is Participating in Psychological Research a Benefit, Burden, or Both for Medically Ill Youth and Their Caregivers? IRB. 2015 Nov-Dec;37(6):1-8. PMID 26783591